CLINICAL TRIAL: NCT07096661
Title: Expert Perspectives on Pain Science Education for Labour and Postpartum Pain: A Delphi Study
Brief Title: Pain Science Education for Labour and Postpartum Pain
Acronym: PNE-DELPHI
Status: Not yet recruiting | Type: Observational
Sponsor: Bournemouth University (Other)
Collaborators: Akdeniz University (Other); Vrije Universiteit Brussel (Other); McMaster University (Other)
Responsible Party: Principal Investigator, Omer Elma, Lecturer, Bournemouth University
Other Study IDs: 61318
Record Dates: First submitted 2025-07-14; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Adults; Female; Labour Pain; Postpartum Pain; Chronic Pain
Keywords: Pain Neuroscience Education; PNE; Postpartum Pain; Natal Pain; Labor Pain; Delphi Study; persistent pain
MeSH Terms: conditions — Labor Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This Delphi study aims to establish expert consensus on the role, content, and delivery of pain science education (PSE) for labour and postpartum pain management. Despite the growing application of PSE in other populations, its use in maternity care remains underexplored. Through a three-round electronic Delphi survey, multidisciplinary experts-including physiotherapists, midwives, gynaecologists, pain specialists, nurses, and psychologists-will contribute their perspectives to guide the development of a structured PSE intervention for future clinical testing.

DETAILED DESCRIPTION:
Labour pain is a critical and complex experience that can significantly influence both immediate and long-term maternal outcomes. Although antenatal education often addresses pain minimally or inconsistently, pain science education (PSE)-which reconceptualizes pain as a biopsychosocial phenomenon-has demonstrated benefits in other clinical contexts, such as chronic pain and musculoskeletal rehabilitation. PSE may reduce fear, enhance coping strategies, and support physiological birth outcomes. However, its integration into maternity care, particularly during labour and postpartum periods, has yet to be defined.

This study employs a three-round electronic Delphi (e-Delphi) methodology to gain consensus on the use of PSE in this context. The Delphi method is ideal for topics where empirical evidence is limited but expert opinion is available. Guided by established best practices including the CREDES (Guidance on Conducting and REporting DElphi Studies) this study ensures methodological rigour and transparency.

Multidisciplinary experts will be purposively recruited internationally via professional networks and social media platforms. To participate, experts must be English-speaking adults with relevant clinical experience or academic contributions in PSE, pain management, or antenatal education. The study will include physiotherapists, midwives, gynaecologists, psychologists, nurses, and pain specialists. Participants will be provided with detailed study information and will give informed consent electronically.

The Delphi process will be conducted in three iterative rounds, allowing experts to respond anonymously to survey items, review aggregate group feedback, and refine their views. This method aims to identify convergence in expert perspectives and clarify the key components of a future PSE intervention for labour and postpartum care. Data will be analysed using NVivo for qualitative responses and SPSS for quantitative analysis.

The outcome of this study will inform the development of a clearly defined, evidence-informed PSE intervention to be tested in future clinical trials. It represents an important step toward improving antenatal education and enhancing pain management during and after childbirth.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Ability to read and write in English
* Professional background as one of the following:

Registered physiotherapist Registered midwife Gynaecologist Pain management specialist Nurses Psychologist

Exclusion Criteria:

* Inability to read or write in English
* Lack of relevant professional background or clinical experience as outlined in the inclusion criteria
* Decline or fail to provide informed consent
* Under 18 years of age

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of 30 multidisciplinary experts recruited internationally, including physiotherapists, midwives, gynaecologists, pain management specialists, nurses, and psychologists. These participants will be selected using purposive sampling to ensure a diverse representation of professional backgrounds and experiences related to pain science education, pain management, and antenatal care.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Expert Consensus on Content of Pain Science Education for Labour and Postpartum | Day 2
  Expert consensus will be assessed using a structured three-round electronic Delphi survey. Survey items will ask participants to rate the importance or relevance of specific pain science education topics and components using a 5-point Likert scale (1 = not important to 5 = essential). Consensus will be defined as ≥70% of participants rating an item as either 4 or 5. Quantitative agreement levels will be calculated per item in SPSS, and qualitative comments will be analysed in NVivo to support interpretation of ratings.
Expert Consensus on Optimal Timing for Delivery of Pain Science Education | Day 2
  Expert consensus on optimal time points for delivering pain science education will be assessed using a structured three-round electronic Delphi survey. Participants will rate each proposed timing option using a 5-point Likert scale (1 = not appropriate to 5 = highly appropriate). Consensus will be defined as ≥70% of experts rating an item as 4 or 5. Quantitative data will be analysed using SPSS.
Expert Consensus on Preferred Delivery Methods for Pain Science Education | Day 2
  Expert agreement on preferred delivery formats for PSE (e.g., individual vs. group sessions, online vs. in-person, specific provider roles) will be assessed via a structured e-Delphi survey. Items will be rated on a 5-point Likert scale (1 = not feasible/effective to 5 = highly feasible/effective). Consensus will be defined as ≥70% of participants selecting 4 or 5. Quantitative data will be analysed in SPSS to determine consensus levels.

SECONDARY OUTCOMES:
Qualitative Insights into Implementation Feasibility and Barriers | Day 3
  Open-ended responses collected during the e-Delphi rounds will be analysed thematically to identify perceived barriers, facilitators, and implementation considerations for integrating PSE into routine antenatal care. Data will be analysed using qualitative content analysis in NVivo, with codes developed inductively and reviewed by multiple researchers to ensure rigour.

CONTACTS AND LOCATIONS:
Locations (1):
- Landsdowne Campus, Bournemouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No